CLINICAL TRIAL: NCT03538470
Title: Clinical Evolution of Patients Suffering From Lower Limb Rheumatological Conditions 6 Months After Spa Treatment
Brief Title: Assessment of the Effect of Spa Treatment on Rheumatological Conditions
Acronym: CONTREXEVILLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SAEML Contrexéville (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 1.3
Record Dates: First submitted 2018-04-17; First posted 2018-05-29 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Knee; Pain, Joint; Lower Back Pain; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia; Low Back Pain; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spa treatment (Experimental): Mineral water cares in Contrexéville thermal cure center, massage, cataplasm.
  Interventions: Other: Spa Treatment

INTERVENTIONS:
Other: Spa Treatment — * Bath with immersion shower
  * Overall penetrating shower
  * Multiple local application cataplasm
  * Individual physiotherapy
  * Mobilisation pool

SUMMARY:
1. Primary outcome measure: measuring the effect of spa treatment in patients suffering from lower limb osteoarthritis or any other lower limb rheumatological condition.

   Percentage of patients with minimum 19,9 mm decrease in pain Visual Analogue Scale (VAS) or WOMAC score (Western Ontario and McMaster Universities Arthritis Index) improvement of at least 9 points (minimal clinically important difference), 6 months after enrollment.

   Secondary outcome measures:
2. Measuring the effect of spa treatment in patients with concomitant chronic lower back pain.

   Percentage of patients presenting clinical benefits according to the EIFEL score, with a decrease of at least 5 points, 6 months after enrollment.
3. Quantitative evaluation of pain. Mean pain VAS comparison between enrollment and 6 months after spa treatment.
4. Quantitative evaluation of WOMAC score. Mean WOMAC score comparison between enrollment and 6 months after spa treatment.
5. Quantitative evaluation of EIFEL score. Mean EIFEL score comparison between enrollment and 6 months after spa treatment.
6. Impact of spa treatment on the patient's metabolism. Height and weight (BMI calculation), blood pressure and heart rate measured at enrollment and throughout the follow-up.
7. 8. Quality of life. 36-Item Short Form (SF 36) and EuroQol 5 Dimensions (EQ5D) questionnaires at enrollment, 3 months and 6 months.

9. Doctor and patient opinion. Semi-quantitative scale collected at enrollment, 3 months and 6 months.

10. Medicine consumption Daily medicine consumption evaluated upon the 72 hours preceding the medical visit at enrollment, 3 months and 6 months.

11. Auto-evaluation of pain VAS pain evaluation by the patient every 6 weeks for a more precise time frame of the treatment's effect.

DETAILED DESCRIPTION:
Osteoarthritis and rheumatic conditions in general are a major public health issue, notably causing chronic pain disorders.

Spa treatments currently play a central role in the non-medical therapeutic arsenal for patients suffering from these rheumatic diseases.

A French study estimated the direct costs generated by osteoarthritis in France up to 1,6 billion euros in 2002, half of which was due to hospital expenses (800 million euros). Osteoarthritis required 13 millions consults and drug expenses of 570 million euros. Compared to 1993, these expenses increased by 156% due to the raise of the number of patients treated (+54%) and of the cost for each patient (+2,5% per year). This study concerned patients with lower limb osteoarthritis, and a significant portion of these expenses were attributable to the disease.

Chronic lower back pain is also a major health issue for its impact on patients' functional capacities as well as for the economic and social costs it generates. This is a frequent condition, it is estimated that 80% of the population will present lower back pain at some point in their life. Furthermore, epidemiological studies show an increase in the prevalence of lower back pain (3,9% in 1992 to 10,2% in 2006 in the American population).

Different well-conducted studies around the impact of spa treatments have led to the recognition of its beneficial outcome on the treatment of chronic lower back pain.

Several controlled, randomized, prospective trials have already evaluated the effect of spa treatment for other main indications claimed by crenotherapy in rheumatology such as hip and hand osteoarthritis, fibromyalgia, rheumatoid polyarthritis, psoriatic arthritis and chronic neck pain.

The THERMARTHROSE study by Forestier demonstrated the efficacy of spa treatments as a rheumatological indication for knee osteoarthritis using the WOMAC questionnaire and VAS pain scale. Following the model of this study, the investigators chose to use the WOMAC and VAS pain scale as the primary endpoints of the investigator's study.

The WOMAC questionnaire was developed by Bellamy in 1988, it is a functional index centered on the locomotor system.

The pain VAS is an auto-evaluation tool derived from visual analogue scales developed in psychiatry to measure patients' well-being. Today, this statistically measurable and reproductible tool is commonly used in clinical trials to monitor the evolution of pain and more precisely to evaluate the impact of a treatment on a given chronic disease such as osteoarthritis. For this study, pain will be measured using pain VAS according to Huskinsson and following methodology as recommended by French health authorities, with one measure.

During clinical studies in thermal environment, spa treatment is a composite entity including the effect of the water itself, but also physiotherapy, rest, education… The spa of Contrexéville wishes to obtain a new rheumatic indication. According to the recommendations of the Academy of Medicine, a prolonged observation of a cohort with repeated measures is required for any spa wishing to acquire the accreditation for a new orientation.

Towards this aim, the investigators wish to undertake a prospective study with repeated measures in order to analyze the evolution of the clinical state of patients with a rheumatic disease on the lower limbs or the rachis, 6 months after receiving a spa treatment in the Contrexéville thermal institute. Since rheumatological treatments at Contrexéville are not covered by health insurance, they will not be billed to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting an indication for rheumatological spa treatment
* Patient with osteoarthritis or other rheumatic disease, located on the lower limbs with or without chronic lower back pain.
* Functional impairment with reduced mobility
* Life expectancy > 6 months
* VAS pain evaluation > 30 mm
* Available for a 6-months follow-up and an 18-days spa treatment
* Affiliation to the French social security system or equivalent
* Patient living within 100 kms of recruitment center

Exclusion Criteria:

* Patient having already underwent a spa treatment for rheumatic indication 6 months within enrollment
* Pregnancy, parturient or breast feeding
* Psychiatric illness or social situation that would preclude study compliance
* Predictable intolerance to thermal treatment (immunodeficiency, advanced cardiopathy, active cancer, active pulmonary tuberculosis, severe renal failure, cirrhosis, advanced dementia and severe mental conditions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of spa treatment on lower limb osteoarthritis | At 6 months
  Percentage of patients with a WOMAC score improvement of 9 or more points and/or with a decrease in VAS of at least 19,9 mm (minimal clinically important difference)

SECONDARY OUTCOMES:
Effect of spa treatment on lower back pain | At 6 months
  Percentage of patients with an EIFEL score decrease of at least 5 points
Quantitative evaluation of pain | At baseline and 6 months
  Comparison of mean VAS (Visual Analogic Scale from 0 to 10) pain scale
Quantitative evaluation of WOMAC | At baseline and 6 months
  Comparison of mean WOMAC questionnaire
Quantitative evaluation of EIFEL | At baseline and 6 months
  Comparison of mean EIFEL questionnaire
Patient BMI | At baseline, 3 and 6 months
  BMI evolution will be recorded (size, weight)
Global quality of life | At baseline, 3 and 6 months
  SF36 (The Short Form (36) Health Survey) questionnaire will be recorded. The SF36 questionnaire includes 36 questions from which eight dimensions and two aggregate scores (the physical dimension and the psychic dimension) are calculated. The correction of the missing data and the different methods of adjustment and calculation of the scores will be carried out according to the procedure recommended by the manual. The scores of the different dimensions range from 0: less good health and 100: the best.
Health quality of life | At baseline, 3 and 6 months
  EQ5D questionnaire will be recorded. EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ5D has 6 items intended to measure general health. The top 5 rate mobility, independence, daily activities, pain / discomfort, and anxiety / depression, and are rated according to 3 values from "No problem" to "Problem" or "Incapacity". This results in an index score. The last item deals with perceived health on the day the questionnaire is filled in and uses a visual analogue scale from 0 (worst) to 100 (best health possible) (Visual Analog Scale Score).
Doctor / patient opinions | At baseline, 3 and 6 months
  Semi-quantitative scale in 7 points collected will be recorded. This is a semi-quantitative evaluation of the effect of the cure on the state of health of the patient by the patient himself and the same questions by the doctor. Responses will be grouped into 3 classes: aggravated / neither aggravated nor improved / improved. The numbers and percentages of each answer will be calculated
Treatment follow-up | At baseline, 3 and 6 months
  Description of treatments consumption by the patient at baseline, 3 and 6 months. To avoid any risk of confusion, drug consumption will be related to daily consumption. Drug use for 72 hours (day before and before the day of visit, day of visit: d-2, d-1, D0)
Self evaluation of pain | With investigator at baseline, 3 and 6 months. Auto evaluation at 1.5 months and 4.5 months.
  Visual Analogic Scale (from 0 to 10) evaluation by patients

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc BOSSON, MD, Study Chair — TIMC-IMAG
Locations (4):
- France (4):
  - Conrozier, Belfort
  - BAUER, Nancy
  - Perrier Cornet, Nancy
  - Jeanmaire, Neufchâteau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Buskila D, Abu-Shakra M, Neumann L, Odes L, Shneider E, Flusser D, Sukenik S. Balneotherapy for fibromyalgia at the Dead Sea. Rheumatol Int. 2001 Apr;20(3):105-8. doi: 10.1007/s002960000085. PMID 11354556
- [Background] Constant F, Collin JF, Guillemin F, Boulange M. Effectiveness of spa therapy in chronic low back pain: a randomized clinical trial. J Rheumatol. 1995 Jul;22(7):1315-20. PMID 7562765
- [Background] Constant F, Guillemin F, Collin JF, Boulange M. Use of spa therapy to improve the quality of life of chronic low back pain patients. Med Care. 1998 Sep;36(9):1309-14. doi: 10.1097/00005650-199809000-00003. PMID 9749654
- [Background] Elkayam O, Ophir J, Brener S, Paran D, Wigler I, Efron D, Even-Paz Z, Politi Y, Yaron M. Immediate and delayed effects of treatment at the Dead Sea in patients with psoriatic arthritis. Rheumatol Int. 2000;19(3):77-82. doi: 10.1007/s002960050107. PMID 10776684
- [Background] Evcik D, Kizilay B, Gokcen E. The effects of balneotherapy on fibromyalgia patients. Rheumatol Int. 2002 Jun;22(2):56-9. doi: 10.1007/s00296-002-0189-8. Epub 2002 Mar 29. PMID 12070676
- [Background] Franke A, Reiner L, Pratzel HG, Franke T, Resch KL. Long-term efficacy of radon spa therapy in rheumatoid arthritis--a randomized, sham-controlled study and follow-up. Rheumatology (Oxford). 2000 Aug;39(8):894-902. doi: 10.1093/rheumatology/39.8.894. PMID 10952746
- [Background] Guillemin F, Constant F, Collin JF, Boulange M. Short and long-term effect of spa therapy in chronic low back pain. Br J Rheumatol. 1994 Feb;33(2):148-51. doi: 10.1093/rheumatology/33.2.148. PMID 8162480
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Konrad K, Tatrai T, Hunka A, Vereckei E, Korondi I. Controlled trial of balneotherapy in treatment of low back pain. Ann Rheum Dis. 1992 Jun;51(6):820-2. doi: 10.1136/ard.51.6.820. PMID 1535495
- [Background] Levy E, Ferme A, Perocheau D, Bono I. [Socioeconomic costs of osteoarthritis in France]. Rev Rhum Ed Fr. 1993 Jul;60(6 Pt 2):63S-67S. French. PMID 8118454
- [Background] Driscoll T, Jacklyn G, Orchard J, Passmore E, Vos T, Freedman G, Lim S, Punnett L. The global burden of occupationally related low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):975-81. doi: 10.1136/annrheumdis-2013-204631. Epub 2014 Mar 24. PMID 24665117
- [Background] Leplege A, Ecosse E, Verdier A, Perneger TV. The French SF-36 Health Survey: translation, cultural adaptation and preliminary psychometric evaluation. J Clin Epidemiol. 1998 Nov;51(11):1013-23. doi: 10.1016/s0895-4356(98)00093-6. PMID 9817119
- [Background] Neumann L, Sukenik S, Bolotin A, Abu-Shakra M, Amir M, Flusser D, Buskila D. The effect of balneotherapy at the Dead Sea on the quality of life of patients with fibromyalgia syndrome. Clin Rheumatol. 2001;20(1):15-9. doi: 10.1007/s100670170097. PMID 11254234
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state. Ann Rheum Dis. 2005 Jan;64(1):34-7. doi: 10.1136/ard.2004.023028. Epub 2004 May 6. PMID 15130902
- [Background] van Tubergen A, Landewe R, van der Heijde D, Hidding A, Wolter N, Asscher M, Falkenbach A, Genth E, The HG, van der Linden S. Combined spa-exercise therapy is effective in patients with ankylosing spondylitis: a randomized controlled trial. Arthritis Rheum. 2001 Oct;45(5):430-8. doi: 10.1002/1529-0131(200110)45:53.0.co;2-f. PMID 11642642
- [Background] Van Tubergen A, Boonen A, Landewe R, Rutten-Van Molken M, Van Der Heijde D, Hidding A, Van Der Linden S. Cost effectiveness of combined spa-exercise therapy in ankylosing spondylitis: a randomized controlled trial. Arthritis Rheum. 2002 Oct 15;47(5):459-67. doi: 10.1002/art.10658. PMID 12382292
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Woodforde JM, Merskey H. Some relationships between subjective measures of pain. J Psychosom Res. 1972 Jun;16(3):173-8. doi: 10.1016/0022-3999(72)90041-4. No abstract available. PMID 5072910
- [Background] Marty M, Courvoisier D, Foltz V, Mahieu G, Demoulin C, Gierasimowicz A, Norberg M, de Goumoens P, Cedraschi C, Rozenberg S, Genevay S; Section Rachis de la Societe Francaise de Rhumatologie. How much does the Dallas Pain Questionnaire score have to improve to indicate that patients with chronic low back pain feel better or well? Eur Spine J. 2016 Jan;25(1):304-309. doi: 10.1007/s00586-015-3957-3. Epub 2015 Apr 23. PMID 25904420
- [Background] Sun SF, Hsu CW, Lin HS, Liou IH, Chen YH, Hung CL. Comparison of Single Intra-Articular Injection of Novel Hyaluronan (HYA-JOINT Plus) with Synvisc-One for Knee Osteoarthritis: A Randomized, Controlled, Double-Blind Trial of Efficacy and Safety. J Bone Joint Surg Am. 2017 Mar 15;99(6):462-471. doi: 10.2106/JBJS.16.00469. PMID 28291178
- [Background] Verhagen AP, de Vet HC, de Bie RA, Kessels AG, Boers M, Knipschild PG. Balneotherapy for rheumatoid arthritis and osteoarthritis. Cochrane Database Syst Rev. 2000;(2):CD000518. doi: 10.1002/14651858.CD000518. PMID 10796385
- [Background] Coste J, Le Parc JM, Berge E, Delecoeuillerie G, Paolaggi JB. [French validation of a disability rating scale for the evaluation of low back pain (EIFEL questionnaire)]. Rev Rhum Ed Fr. 1993 May;60(5):335-41. French. PMID 8167640
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Grotle M, Brox JI, Vollestad NK. Concurrent comparison of responsiveness in pain and functional status measurements used for patients with low back pain. Spine (Phila Pa 1976). 2004 Nov 1;29(21):E492-501. doi: 10.1097/01.brs.0000143664.02702.0b. PMID 15507789
- [Background] Maughan EF, Lewis JS. Outcome measures in chronic low back pain. Eur Spine J. 2010 Sep;19(9):1484-94. doi: 10.1007/s00586-010-1353-6. Epub 2010 Apr 17. PMID 20397032
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131